CLINICAL TRIAL: NCT01792752
Title: Enhanced Access to HIV Care for Drug Users in San Juan, Puerto Rico
Acronym: Proyecto PACTo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: University of Puerto Rico (Other); Iniciativa Comunitaria de Investigacion (Unknown); Puerto Rico Department of Health (Unknown); University of Miami (Other); Weill Medical College of Cornell University (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Lisa Metsch, Stephen Smith Professor and Chair of Sociomedical Sciences Department, Columbia University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AAAK8805; 1R01DA035280-01 (NIH)
Record Dates: First submitted 2013-02-08; First posted 2013-02-15 (Estimated); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: HIV; AIDS; Substance Abuse
Keywords: HIV/AIDS; Drug Users; Puerto Rico
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Substance-Related Disorders; Drug Misuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced HIV Care Access and Retention Intervention (Experimental): Through the Enhanced HIV Care Access and Retention Intervention, the five neighborhoods will receive the 4 components of the intervention: 1) HIV Testing Campaign; 2) Treatment Re-engagement Campaign; 3) Patient Navigator Linkage to Care and Substance Abuse Treatment Team; and 4) Mobile Care Clinic. The neighborhoods will receive the intervention at different times throughout the study period, but once the intervention is initiated in a neighborhood it will continue being implemented in that neighborhood until the end of the study period.
  Interventions: Behavioral: Enhanced HIV Care Access and Retention Intervention; Behavioral: HIV Testing Campaign; Behavioral: Treatment Re-engagement Campaign; Behavioral: Patient Navigator Linkage to Care and Substance Abuse Treatment Team; Behavioral: Mobile Care Clinic
- Control / Neighborhood(s) not receiving the intervention (No Intervention): The neighborhood(s) not receiving the intervention will act as a control while the intervention is initiated and implemented in other neighborhoods. All neighborhoods will receive the intervention but at different times throughout the study period. Once the intervention is initiated in a neighborhood, that neighborhood will continue receiving the intervention until the end of the study period.

INTERVENTIONS:
Behavioral: Enhanced HIV Care Access and Retention Intervention — Through the Enhanced HIV Care Access and Retention Intervention, the five neighborhoods will receive the 4 components of the intervention: 1) HIV Testing Campaign; 2) Treatment Re-engagement Campaign; 3) Patient Navigator Linkage to Care and Substance Abuse Treatment Team; and 4) Mobile Care Clinic. In addition to these intervention components, study participants will receive screening and access to treatment for other physical and mental co-morbidities, general primary health care, and social/psychosocial services addressing unstable housing, food insecurity, interpersonal violence, legal issues. All HIV-positive IDUs identified either through the HIV Testing Campaign or the Treatment Re-engagement Campaign will be enrolled in the HIV Care Cohort. The HIV Care Cohort will be comprised of the HIV-positive injectors who are receiving direct services in the Mobile Care Clinic. The 4 intervention components are detailed below:
  Arms: Enhanced HIV Care Access and Retention Intervention
Behavioral: HIV Testing Campaign — When the intervention is initiated in a neighborhood, HIV rapid testing will begin and continue in a particular neighborhood from the time that the neighborhood's intervention begins until the end of the study period. Anyone testing HIV positive will be seen and counseled by a member of the Patient Navigator Team.
  Arms: Enhanced HIV Care Access and Retention Intervention
Behavioral: Treatment Re-engagement Campaign — Simultaneously with the introduction of the HIV Testing Campaign, a patient navigator team will approach HIV-positive IDUs identified as not having seen their HIV care provider in the last 6 months. In addition, known HIV-positive IDUs within the designated neighborhoods will be approached for service enrollment and meet with a patient navigator.
  Arms: Enhanced HIV Care Access and Retention Intervention
Behavioral: Patient Navigator Linkage to Care and Substance Abuse Treatment Team — The patient navigator team will provide informational support to the HIV-positive injectors, motivate them to attend HIV care visits and engage in substance abuse treatment, encourage their use of and adherence to antiretroviral therapies, and work with them to overcome any barriers to attendance at HIV care visits and substance abuse treatment. All clients of the patient navigator will become part of the HIV Care Cohort; they will have been identified either in the HIV Testing Campaign or the Treatment Re-Engagement Campaign.
  Arms: Enhanced HIV Care Access and Retention Intervention
Behavioral: Mobile Care Clinic — Participants who choose to receive services in the study mobile HIV care clinic will receive an initial appointment and the patient navigator will ensure that the client attends it. At the initial visit, clients will have a medical history taken, be examined and have blood drawn to measure CD4 and viral load. The mobile care clinic doctor will also prescribe medications for the client at the subsequent visit which will be scheduled as soon as lab results are available and interpreted, approximately one week later. The mobile HIV care clinic van will provide health services to the general IDU population within each intervention neighborhood to avoid any stigmatization of the HIV positive clients.
  Arms: Enhanced HIV Care Access and Retention Intervention

SUMMARY:
The overall goal of this project is to implement and evaluate a community-level, structured approach to enhance HIV care access and retention for drug users in San Juan, Puerto Rico. The "Enhanced HIV Care Access and Retention Intervention" will: 1) identify drug users living with HIV who either do not know their HIV status and/or are not engaged in HIV care; 2) provide direct HIV care services through a mobile health van; and 3) support identified HIV-infected drug users with patient navigators to enhance their ability to engage in HIV care and substance abuse treatment, to initiate antiretroviral therapy, and maintain adherence to their treatment regimens. The structural enhanced care approach will be evaluated through a randomized roll-out design, a refinement of the stepped-wedge design. The community-level success of the intervention will be assessed by evaluating virologic suppression (primary biological outcome), increased attendance to HIV care visits, uptake of antiretroviral therapy, adherence to HIV treatment regimens, and decreased substance use (as secondary behavioral outcomes) in an independent cohort of HIV-positive individuals drawn from each of the neighborhoods included in the intervention. The investigators will also evaluate the implementation process and cost of the enhanced care approach including implications for cost-effectiveness, feasibility of expansion, and sustainability.

DETAILED DESCRIPTION:
Recent scientific advances demonstrate that for people living with HIV, antiretroviral therapy (ART) is the most effective strategy to improve immune function, reduce morbidity, improve quality of life, prolong survival, and prevent HIV transmission. Translating this knowledge into practice, however, requires prompt diagnosis and linkage to care, entry into care with timely ART initiation, and engagement in care, support for ART adherence, and retention to promote durable viral suppression. Addressing failures in this cascade of care, often referred to as the "Seek, Test, Treat, and Retain (STTR)" paradigm, has become a major part of the National HIV/AIDS strategy in the United States. To date, much of the research and discussion surrounding this strategy has focused on expanding HIV testing to improve the early identification of new cases. There has been less attention focused on linkage to, engagement in, and retention in care. Specifically, little attention has focused on identifying HIV-positive individuals who, despite being aware of their diagnosis, have never been in HIV care, are intermittent users of care, or have dropped out of care.

HIV-infected injection drug users (IDUs) are a particularly difficult subpopulation to link to and retain in HIV care. They face a myriad of challenges that can impede retention in care including substance use disorders (both alcohol and drugs), mental health problems and poverty-related issues such as unstable housing and food insecurity. If IDUs adhere to their treatment regimens, however, studies have demonstrated they realize similar survival benefits from antiretroviral therapy as persons without a history of injection drug use. In contrast to the majority of communities in the U.S., in Puerto Rico, drug use, particularly injection drug use, continues to fuel a fast-growing HIV epidemic. Puerto Rico has an estimated incidence rate of 45 HIV cases per 100,000 population, twice the rate for the 50 U.S. states, and almost 40% of new infections are associated with injection drug use. In contrast, only 12% of new infections in the 50 U.S. states are among IDUs.

The overall goal of this project is to implement and evaluate a community-level, structured enhanced approach, the Enhanced HIV Care Access and Retention Intervention, for substance users in San Juan, Puerto Rico. It will bring HIV care directly to five San Juan zones in which a high proportion of HIV-infected substance users reside. The significance of the study is threefold.f care, or have dropped out of care.

ELIGIBILITY:
HIV Testing Campaign

Inclusion Criteria:

1. be 18 years of age or older
2. report having injected drugs (opioid or stimulants) at least once in the past 30 days
3. provide written informed consent

HIV Care Cohort

Inclusion Criteria:

1. be 18 years of age or older
2. test HIV-seropositive through rapid testing (confirmed with Western Blot or immunofluorescence assay)
3. report having injected drugs more than once per week for the past 30 days
4. self-report that they have not been in HIV care for the past 6 months
5. agree to have their blood drawn for CD4 and HIV plasma RNA testing
6. live in one of the San Juan neighborhoods targeted for intervention
7. provide basic contact information for follow-up
8. sign a HIPAA Authorization/medical record release form
9. provide written informed consent

Assessment Cohort

Inclusion Criteria:

1. be 18 years of age or older
2. test HIV-seropositive through rapid testing (confirmed with Western Blot or immunofluorescence assay)
3. report having injected drugs more than once per week for the past 30 days
4. self-report that they have not been in HIV care for the past 6 months
5. agree to have their blood drawn for CD4 and HIV plasma RNA testing
6. live in one of the San Juan neighborhoods targeted for intervention
7. provide basic contact information for follow-up
8. sign a HIPAA Authorization/medical record release form
9. provide written informed consent

Exclusion Criteria (for all study components mentioned above):

1. do not meet any one or more of the above-described inclusion criteria
2. have significant cognitive or developmental impairment to the extent that they are unable to provide informed consent
3. are terminated via Site PI decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2082 (Actual)
Dates: Start 2013-12-20 (Actual); Primary Completion 2020-08 (Actual); Study Completion 2021-07 (Actual)

PRIMARY OUTCOMES:
HIV Virologic Suppression | Every 6 months for up to 36 months
  Assessment of success of the intervention will be measured by testing whether there is a significant change in virologic suppression associated with the intervention.

SECONDARY OUTCOMES:
Increasing HIV care visit attendance | Every 6 months for up to 36 months
Uptake of antiretroviral therapy | Every 6 months for up to 36 months
Adherence to HIV treatment regimens | Every 6 months for up to 36 months
Decreasing substance use | Every 6 months for up to 36 months
Consistency of enrollment in the intervention and receipt of intervention services across neighborhoods over time | 36 months
Cost of delivering the intervention and of other medical services received | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Metsch, Ph.D., Principal Investigator — Columbia University; Jorge Santana, M.D., Principal Investigator — University of Puerto Rico Medical Sciences Campus; Sandra Miranda De Leon, M.P.H., Principal Investigator — Puerto Rico Department of Health; Daniel Feaster, Ph.D., Principal Investigator — University of Miami; Bruce Schackman, Ph.D., Principal Investigator — Joan & Sanford I. Weill Medical College of Cornell University; Glenda Davila, M.D., Principal Investigator — Iniciativa Comunitaria de Investigacion, Inc.; Lauren K. Gooden, Ph.D, Study Director — Columbia University
Locations (2):
- Puerto Rico (2):
  - Puerto Rico Department of Health, Rio Piedras
  - Iniciativa Comunitaria de Investigacion, Inc., San Juan